CLINICAL TRIAL: NCT01343615
Title: Hemodynamic Alterations in Middle Cerebral Artery and Intraoperative Microemboli During Carotid Endarterectomy and Angioplasty
Brief Title: Study of Blood Flow Changes and Microemboli During Carotid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Hemodynamic alterations in middle cerebral artery and intraoperative microemboli during carotid endarterectomy and angioplasty, Unicamp
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MES2011
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Carotid Endarterectomy; Percutaneous Transluminal Angioplasty; Cognitive Aspects; Diffusion Weighted MRI
MeSH Terms: interventions — Endarterectomy, Carotid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- carotid stenting (Active Comparator)
  Interventions: Procedure: carotid stenting
- carotid endarterectomy (Active Comparator)
  Interventions: Procedure: carotid endarterectomy

INTERVENTIONS:
Procedure: carotid stenting — A group of patients will be operated by endovascular technique. Then will be analyzed and compared with the other group in relation to clinical and radiological criteria, emphasizing the cognitive aspects.
  Arms: carotid stenting
Procedure: carotid endarterectomy — A group of patients will be operated by open technique. Then will be analyzed and compared with the other group in relation to clinical and radiological criteria, emphasizing the cognitive aspects
  Arms: carotid endarterectomy

SUMMARY:
The purpose of this study is to determine the clinical and radiologic implications of the intraoperative microemboli during carotid revascularization.

ELIGIBILITY:
Inclusion Criteria:

* acoustic window for transcranial Doppler
* surgical criteria proposed by the NASCET and ACAS studies
* postoperative follow-up for at least six months
* patient consent

Exclusion Criteria:

* carotid restenosis
* combined surgery
* emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-01 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic alterations in middle cerebral artery and intraoperative microemboli during carotid endarterectomy and angioplasty | 6 months
  The blood flow velocity of the middle cerebral artery will be measured in cm / s and the number of microemboli will be represented by the number of microemboli signals measured by transcranial Doppler ultrasound.
Number of ischemic areas detected by magnetic resonance | 6 months
Neuropsychological changes | 6 months
  Neuropsychological alterations will be assessed through cognitive tests, which generate scores. It will be used: Mini Mental State Examination, Rey's Auditory-Verbal Learning Test, Copy and evocation of Rey's Complex Figure, Weschsler's Immediate Memory Test (direct and indirect digit span ), Lexical and Categorical Verbal Fluency, Stroop Test, Visuospatial Perception Test of Luria's Neuropsychological Investigation, Trail Making Test A e B, Boston Naming Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clínicas da Unicamp, Campinas, São Paulo, Brazil